CLINICAL TRIAL: NCT01679275
Title: Longitudinal Pre-operative Measurements of Cerebral Oxygenation Using Near Infrared Spectroscopy in Neonates With Congenital Heart Disease.
Brief Title: Pre-operative Cerebral Oxygenation in Neonates With Congenital Heart Disease
Acronym: CHD-NIRS
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S54683
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2023-01-30 (Actual); Status verified 2018-05

CONDITIONS: Heart Defects, Congenital
Keywords: Heart Defects, congenital; Patient Monitoring; Infant, Newborn; Physiology
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- measuring cerebral oxygenation: NIRS: Measurement of cerebral oxygenation using Near Infrared Spectroscopy (NIRS) during the pre-operative phase in neonates with congenital heart disease.
  Interventions: Other: measuring cerebral oxygenation

INTERVENTIONS:
Other: measuring cerebral oxygenation

SUMMARY:
Congenital heart disease with need for early surgery in newborns is associated with an increased incidence in global impairment in development. The causes of these late adverse neurologic outcomes are multifactoral and include both fixed (or patient-specific factors) and modifiable factors. They relate to both the mechanism of central nervous system injury associated with congenital heart disease and its treatment. Measuring cerebral oxygenation is a promising non-invasive way of cerebral monitoring in a neonatal intensive care unit. The importance of cerebral monitoring in neonates with congenital heart problems at risk of developing neurological complications is increasingly recognized. In this way the most vulnerable moments for the newborn brain can be detected and ,if possible, lead to change in (timing of) treatment.

ELIGIBILITY:
Inclusion Criteria:

* neonates with admission on neonatal intensive care unit with congenital heart disease.

Exclusion Criteria:

* No informed consent. (for the long term neurodevelopmental FU)
* no cerebral oxygen saturation in the first 3 day's of life
* gestational age < 37 weeks

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants with congenital heart defect
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Neurodevelopmental follow up at 24 months | 24 months
  Neurodevelopmental assessment at 24 months using Bayley scales of infant development II

SECONDARY OUTCOMES:
cerebrovascular changes in the transitional phase | first 3 days of life
  Cerebral oxygen saturation and autoregulatory capacity
Association of cerebrovascular changes with short term outcome | time frame of 1 admission
  short term outcome defined as cerebral ultrasound abnormalities at admission and discharge, ICU stay, hospital stay and mortality before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Thewissen, MD, Principal Investigator — UZ Leuven
Locations (1):
- Neonatal Intensive Care Unit UZLeuven, Leuven, Vlaams Brabant, Belgium